CLINICAL TRIAL: NCT04220931
Title: Intrapapillary Botulinum Toxin Injection for PREvention of Post-surgical PAncREactic Fistula
Acronym: PREPARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P170913J
Record Dates: First submitted 2019-12-20; First posted 2020-01-07 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Distal Pancreatectomy; Postoperative Pancreatic Fistula
Keywords: distal pancreatectomy
MeSH Terms: interventions — Botulinum Toxins

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- botulinum toxin injection (Experimental): Injection of Botulinum toxin A 100 UI, single dose administration, in the major papilla, in the Oddi sphincter, during upper gastrointestinal endoscopy.
  The endoscopic procedure will be performed under unconscious sedation with intravenous injection of propofol by an anesthesiologist.
  Interventions: Drug: botulinum toxin injection
- standard care (No Intervention): standard care (no endoscopy)

INTERVENTIONS:
Drug: botulinum toxin injection — injection of Botulinum toxin A 100 UI, single dose administration, in the major papilla, in the Oddi sphincter, during upper gastrointestinal endoscopy.
  Arms: botulinum toxin injection

SUMMARY:
Surgery is required for the treatment of many pancreatic conditions, either malignant or benign. Mortality of pancreatic surgery can be up to 3% even in expert centers. Morbidity is high, postoperative pancreatic fistula (POPF) being the main postoperative complication. In its current definition (drain output of any measurable fluid >= postoperative day 3 with amylase content >3 times the serum amylase activity and with clinical consequence), the incidence of postoperative PF is between 15 and 30 %. Most POPF resolve spontaneously but when refractory POPF occurs, it may lead to severe complications. POPF severity is graded as follows: grade B in case of change in medical management: infection without organ failure, specific medication (total parenteral nutrition, somatostatin analogs, antibiotics), persistent drainage > 3 weeks, angiographic procedure for bleeding, prolonged hospital stay; grade C in case of reoperation or PF-related organ failure or death.

No specific prophylactic treatment of POPF is currently recommended by clinical guidelines. In clinical research, many prophylactic strategies have been attempted with partial efficacy. Endoscopic pancreatic sphincterotomy with plastic stent placement is effective in pre-and postoperative management of pancreatic fistula but with the need of a highly competent interventional endoscopist. Intrapapillary botulinum toxin injection is believed to induce relaxation of the pancreatic sphincter, leading to a " pharmacological " pancreatic sphincterotomy without any morbidity.

A recent phase I/II prospective study has shown promising results in this indication, with no clinically relevant pancreatic fistula when botulinum toxin was injected. Based on this observation we hypothesize that intrapapillary botulinum toxin injection during an endoscopic procedure before surgery could be effective for the prevention of post-surgical pancreatic fistula

DETAILED DESCRIPTION:
Surgery is required for the treatment of many pancreatic conditions, either malignant or benign. Mortality of pancreatic surgery can be up to 3% even in expert centers. Morbidity is high, postoperative pancreatic fistula (POPF) being the main postoperative complication. In its current definition (drain output of any measurable fluid >= postoperative day 3 with amylase content >3 times the serum amylase activity and with clinical consequence), the incidence of postoperative PF is between 15 and 30 %. Most POPF resolve spontaneously but when refractory POPF occurs, it may lead to severe complications. POPF severity is graded as follows: grade B in case of change in medical management: infection without organ failure, specific medication (total parenteral nutrition, somatostatin analogs, antibiotics), persistent drainage > 3 weeks, angiographic procedure for bleeding, prolonged hospital stay; grade C in case of reoperation or PF-related organ failure or death.

No specific prophylactic treatment of POPF is currently recommended by clinical guidelines. In clinical research, many prophylactic strategies have been attempted with partial efficacy. Endoscopic pancreatic sphincterotomy with plastic stent placement is effective in pre-and postoperative management of pancreatic fistula but with the need of a highly competent interventional endoscopist. Intrapapillary botulinum toxin injection is believed to induce relaxation of the pancreatic sphincter, leading to a " pharmacological " pancreatic sphincterotomy without any morbidity.

A recent phase I/II prospective study has shown promising results in this indication, with no clinically relevant pancreatic fistula when botulinum toxin was injected. Based on this observation we hypothesize that intrapapillary botulinum toxin injection during an endoscopic procedure before surgery could be effective for the prevention of post-surgical pancreatic fistula

This study will be a prospective, multicentric, phase III, superiority, controlled, randomized (1:1), open-label, clinical trial with two parallel arms (intrapapillary botulinum toxin versus standard care), using a PROBE (Prospective Randomized Open Blinded End-point) methodology.

Patients with scheduled distal pancreatectomy for any indication

Sources of funding for the trial : French Ministry supports this study by PHRC-N 2017.

The botulinum toxin provides by MERZ France (producer of Xeomin)

ELIGIBILITY:
Inclusion Criteria:

* Patients with scheduled distal pancreatectomy for any indication: open or laparoscopic distal pancreatectomy with or without splenectomy
* Age ≥ 18years

Exclusion Criteria:

* History of myasthenia gravis or Eaton-Lambert syndrome
* Inflammatory myositis <2 years or preexisting motor neuron disease or neuropathies
* ASA score > III
* Pregnancy or lactation
* Altered anatomy of the duodenum and/or the major papilla (prior surgery, prior endoscopic sphincterotomy)
* Scheduled pancreaticoduodenectomy (Whipple procedure)
* Scheduled total pancreatectomy
* Scheduled central pancreatectomy
* Scheduled pancreatic enucleation
* Calcified chronic pancreatitis (suspected on preoperative cross-sectional imaging)
* Pancreas divisum (suspected on preoperative cross-sectional imaging)
* Toxin botulinum contraindications (hypersensitivity to albumin or to saccharose, infection or inflammation at the injection site concerned, generalized muscle weakness)
* Preoperative administration of somatostatin analogs: for long-acting somatostatin analogs, a 1-month washout period is necessary; for short-acting somatostatin analogs, a 24-hours washout period is necessary
* Any kind of surgical method to reinforce the pancreatic stump:
* Use of a bioabsorbable patch
* Use of fibrin glue
* Use of a ligament patch
* Tutorship, trusteeship
* Concurrent participation in other experimental trials
* Not Affiliation to the French social security
* Not Ability to give their consent and not written informed consent
* Distal pancreatectomy extended to neighbouring organs (except spleen and gallbladder) or to the vessels (celiac axis, portal vein)

Secondary exclusion criteria: patients who did not have the planned surgery in less than 4 weeks after the botulinum toxin injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
number of postoperative pancreatic fistula | 3 months
  Clinically relevant POPF (grade B and C) in the 3 months after Distal Pancreatectomy

SECONDARY OUTCOMES:
number of postoperative pancreatic fistulas grade B | 3 months
  Grade of postoperative pancreatic fistulas B based on the ISGPF 2016 update
number of postoperative pancreatic fistulas grade C | 3 months
  Grade of postoperative pancreatic fistulas C based on the ISGPF 2016 update
Quantity of Biochemical leak after surgery | 3 months
  Biochemical leak after surgery
number of Postoperative complications | 3 months
  Postoperative complications :
  * intra-abdominal fluid collection
  * delayed gastric emptying
  * hemorrhage
  * pancreatitis
  * wound infection
  * other infectious complication
CLAVIEN-DINDO classification for post-surgical morbidity | 3 months
  CLAVIEN-DINDO classification for post-surgical morbidity
Number of hospital days | 3 months
  Health economics endpoints : duration of hospital stay
Number of hospital readmissions | 3 months
  Health economics endpoints : hospital readmissions
Number of transfer to intensive care unit and the duration of these stays | 3 months
  Health economics endpoints : transfer to intensive care unit and the duration of these stays
Number of fistularelated postoperative invasive procedures | 3 months
  Health economics endpoints : fistularelated postoperative invasive procedures
overall costs of hospitalization | 3 months
  Health economics endpoints : overall costs
Quality of life EQ-5D-5L questionnaire | 3 months
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state : LEVEL 1: indicating no problem LEVEL 2: indicating slight problems LEVEL 3: indicating moderate problems LEVEL 4: indicating severe problems LEVEL 5: indicating unable to/extreme problems
Number of sides effects (complications) related to the endoscopic botulinum toxin injection | 3 months
  number of sides effects (complications) related to the endoscopic botulinum toxin injection

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Prat, prof, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- PRAT, Clichy, France